CLINICAL TRIAL: NCT05844527
Title: Safety and Efficacy of MRG-001 in Wound Healing and Scar Appearance in Pre-Abdominoplasty Surgical Excisions
Brief Title: Safety and Efficacy of MRG-001 in Wound Healing in Abdominoplasty Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedRegen LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRG2023WH
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Wound of Skin; Abdominal Wound
Keywords: Abdominoplasty; Surgical Excision; Wound Healing; MRG-001; Scar Formation
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRG-001 (Experimental): MRG-001 will be administered subcutaneously at 0.01 mL/kg bodyweight 3 times per week for 3 weeks.
  Interventions: Drug: MRG-001
- Saline (Placebo Comparator): Placebo will be administered subcutaneously at 0.01 mL/kg bodyweight 3 times per week for 3 weeks.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: MRG-001 — MRG-001 is a novel fixed-dose drug combination administered subcutaneously to mobilize stem cells and immunomodulatory cells to the wound to accelerate healing.
  Arms: MRG-001
Drug: Saline — Sterile saline will serve as placebo treatment.
  Arms: Saline

SUMMARY:
Surgical excisions are one of the most frequent cutaneous wounds. This study will compare the safety and preliminary efficacy of a novel fixed-dose combination drug MRG-001 in pre-abdominoplasty surgical excisions and scar appearance in subjects undergoing elective abdominoplasty.

DETAILED DESCRIPTION:
Subjects will undergo surgical excisions in the abdominoplasty area and will be treated with MRG-001 or placebo for 3 weeks. After 6 weeks, the excision area is harvested for analysis and the study is terminated and the abdominoplasty is performed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent (which includes the Photographic Release Form and HIPAA) prior to performing any of the Screening Visit procedures.
2. Outpatient, males and females between 18 to 55 years of age, inclusive, at the time of signing the ICF. Female subjects of childbearing potential must have a negative serum pregnancy test at Visit 1a (Study Part A) and 1b (Study Part B) and practice a reliable method of contraception throughout the study.
3. Seeking or scheduled for standard elective abdominoplasty.
4. Willing to undergo directed excisions under local anesthesia and follow-up prior abdominoplasty and to undergo all follow-up visits after abdominoplasty surgery.
5. Nonsmokers (or other nicotine use) as determined by history (no nicotine use over the past 6 months) and by urine cotinine concentration (< 200 ng/mL) at the Screening Visit and prior to admission.
6. Generally, in good health with no clinically significant abnormalities as determined by medical, history, physical examination, 12-lead ECG and clinical laboratory tests.
7. The following applies to female subjects of childbearing potential:

   • Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (hormonal contraception, abstinence, diaphragm with spermicide, condom with spermicide or intrauterine device) from the Screening Visit until the End-of-study Visit.
8. Body mass index (BMI) between 25 and 35.0 kg/m2, inclusive, at the Screening Visit.
9. Men must be willing to use double-barrier contraception from enrollment until 8 weeks after the last dose of the study drug, if not abstinent.

Exclusion Criteria:

1. Participation in any other clinical trial of an experimental treatment or used an investigational drug within the past 30 days.
2. Subject has a clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, hematological or psychiatric disorder(s) as determined by the Principal Investigator or designee.
3. History of diabetes mellitus or an HbA1C greater than 5.7 percent.
4. History of prior abdominal surgery or abdominal liposuction, cryolipolysis, focused ultrasound or other fat reduction procedures in or near the anterior abdomen within 12 months prior to screening.
5. History of poor or delayed wound healing such as prior wound dehiscence, chronic wound or leg ulcer.
6. History of or evidence of a genetic collagen disorder such as Ehlers-Danlos Syndrome.
7. Operating Physician is unable to design an abdominoplasty incision area of at least 25 cm wide by 12 cm tall at the center of the fusiform.
8. The presence of any abnormality of the skin within the area of the proposed abdominoplasty that, in the opinion of the PI, could interfere with the excision process or grading of the resultant surgical scar (e.g., striae gravidarum, striae distensae, excessive nevi, numerous seborrheic keratoses, tattoos, etc.).
9. History of splenectomy or splenomegaly (spleen weighing >750 g).
10. Currently taking immunomodulating drugs (e.g, interferons, interleukin, JAK1/2 inhibitors/corticosteroids).
11. Female subjects who are pregnant or breastfeeding or planning to breastfeed at any time through 90 days after last dose of IP.
12. History of alcohol and/or illicit drug abuse within 2 years of entry.
13. History of hypersensitivity to MRG-001's components (tacrolimus or plerixafor) or hypersensitivity or intolerance to local anesthetics.
14. Any personal, familial, employment or financial situation that could impede the subject's ability to attend all study visits and successfully complete the entire clinical study.
15. Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study.
16. Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.
17. Subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., vulnerable populations, persons in detention, minors and those incapable of giving consent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the preliminary effectiveness of MRG-001 treatment on tensile strength of the scars. The difference in Newton force will be compared between saline and MRG-001. | Week -6 to 0

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of MRG-001 treatment compared to placebo controls. The number of (serious) adverse events will be compared between MRG-001 and placebo | Week -6 to 0
Evaluate the pharmacokinetics of MRG-001 (plerixafor and tacrolimus) in patients with wounds. The following parameters will be assessed: Maximum concentration, trough levels, Minimum concentrations, Clearance and half-life. | Week -6 to 0
Evaluate the pharmacodynamics of wound healing with MRG-001 treatment by measuring the presence of stem cells and immune cells in the peripheral blood and granulation tissue compared to placebo controls. | Week -6 to 0
Assess the time to full re-epithelization of the wounds assessed by digital photography by three independent plastic surgeons. | Week -6 to 0
Assess the scar appearance by the modified POSAS (PI & Patient) at 6 weeks. | Week -6 to 0
Assess the difference in VAS pain scores. | Week -6 to 0
Incidence of wound infection requiring antibiotic therapy within 28 days after excision. | Week -6 to 0
Assess the effect of MRG-001 on the histological presence of stem cells and immunoregulatory cells in the scars. The number of CD133+, CD34+ FOXP3+, Macrophages will be compared between MRG-001 and placebo in the wound area. | Week -6 to 0

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Galiano, MD FACS, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No